CLINICAL TRIAL: NCT06491524
Title: Disposable 7.5Fr Electronic Flexible Ureteroscope Combined 10Fr Ureteral Access Sheath for Treatment of Renal Stone <2cm
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ningbo No. 1 Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-R022
Record Dates: First submitted 2022-11-23; First posted 2024-07-09 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2022-12

CONDITIONS: Ureteroscopy; Urolithiasis
Keywords: flexible ureteroscope; ureteral guide sheath
MeSH Terms: conditions — Urolithiasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 7.5Fr flexible ureteroscope combined 10Fr ureteral access sheath (Experimental): Using disposable 7.5Fr electronic flexible ureteroscope combined 10Fr ureteral access sheath to treat renal stone <2cm
  Interventions: Device: Using disposable 7.5Fr electronic flexible ureteroscope combined 10Fr ureteral access sheath to treat renal stone <2cm

INTERVENTIONS:
Device: Using disposable 7.5Fr electronic flexible ureteroscope combined 10Fr ureteral access sheath to treat renal stone <2cm — Using disposable 7.5Fr electronic flexible ureteroscope combined 10Fr ureteral access sheath to treat renal stone <2cm

SUMMARY:
Observation efficacy and safety of disposable f7.5 electronic flexible ureteroscope combined f10 ureteral guide sheath for treatment of renal stone <2cm.

DETAILED DESCRIPTION:
Using disposable 7.5Fr electronic flexible ureteroscope combined 10Fr ureteral guide sheath to treat renal stone <2cm, and investigating its efficacy and safety.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with kidney stones less than 2cm who choose to perform "Flexible ureteroscopic holmium laser lithotripsy";
2. Over 18 years old, male or female;
3. No hydronephrosis or mild to moderate hydronephrosis (collection system separation is less than 2cm);
4. The subject has no mental illness or language dysfunction, can understand the situation of this study and has signed an informed consent form, and is estimated to be able to cooperate with the completion of the entire study;
5. No urinary tract infection or no clinical manifestations of urinary tract infection;
6. Patients with urinary tract infection, negative urine culture, and no fever need to undergo antibiotic treatment for more than 3 days; urinary routine examination suggests urinary tract infection, positive urine culture, and patients without fever need to undergo antibiotic treatment for more than 7 days, till the urine culture turns negative.

Exclusion Criteria:

1. Patients with a previous history of ureteral stenosis or who have undergone open, laparoscopic ureteral, nephrectomy and lithotripsy;
2. Fever or urinary tract infection is not treated according to the inclusion criteira;
3. Pregnant women and women's menstrual periods;
4. Cannot tolerate anaesthesia or surgery due to serious systemic diseases, heart disease, lung insufficiency and failure of important organs;
5. Anatomical malformations such as polycystic kidneys, horseshoe kidneys, and ectopic kidneys;
6. Patients with high suspicion of ureteral stenosis or diseases that are considered unsuitable to participate in this clinical study;
7. Patients indwelling double J stent preoperatively;
8. Patients who need bilateral upper urinary tract surgery at the same time.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2022-04-20 (Actual); Primary Completion 2023-10-06 (Actual); Study Completion 2023-10-28 (Actual)

PRIMARY OUTCOMES:
Success rate of Accessing | 1 day
  success rate of UAS placement (SRUP)

SECONDARY OUTCOMES:
Evaluation of intraoperative ureteral injury | 1 day
  Evaluation of intraoperative ureteral injury according to the standards proposed by Traxer et. al.
Stone free rate | 1 and 30 days
  stone free rate (SFR)
overactive bladder symptom score (OABSS) | 1 month
  Overactive bladder symptom score (OABSS) before and after the operation
Quality of life (QOL) questionnaire | 1 month
  Quality of life (QOL) before and after the operation

CONTACTS AND LOCATIONS:
Overall Officials: Li Fang, Doctor, Principal Investigator — Urology of NIngbo First Hospital
Locations (1):
- Ningbo First hospital, Ningbo, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No